CLINICAL TRIAL: NCT06208410
Title: A Clinical Study of JS105 in Combination With Other Anti-tumor Therapies in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study of JS105 in Combination With Other Anti-tumor Therapies in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Risen (Suzhou) Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS105-002-Ib/II
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Fulvestrant; toripalimab; Paclitaxel; Injections; fluzoparib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm A:JS105+Fulvestrant Injection (Experimental): JS105 administered orally, Fulvestrant intramuscularly
  Interventions: Drug: JS105; Drug: Fulvestrant injection
- Arm B:JS105+Fulvestrant Injection+Dalpiciclib Isetionate Tablets (Experimental): JS105 administered orally, Dalpiciclib administered orally, Fulvestrant intramuscularly
  Interventions: Drug: JS105; Drug: Fulvestrant injection; Drug: Dalpiciclib Isetionate Tablets
- Arm C:JS105+Toripalimab Injection (Experimental): JS105 administered orally, Toripalimab intravenous infusion
  Interventions: Drug: JS105; Drug: Toripalimab Injection
- Arm D:JS105+Paclitaxel for Injection (Albumin Bound) (Experimental): JS105 administered orally, Paclitaxel (Albumin Bound) intravenous infusion
  Interventions: Drug: JS105; Drug: Paclitaxel for Injection (Albumin Bound)
- Arm E:JS105+Fluzoparib Capsules (Experimental): JS105 administered orally, Fluzoparib administered orally
  Interventions: Drug: JS105; Drug: Fluzoparib Capsules
- Arm F:JS105+Pyrotinib Maleate Tablets+Capecitabine Tablets (Experimental): JS105 administered orally, Pyrotinib administered orally,Capecitabine administered orally
  Interventions: Drug: JS105; Drug: Pyrotinib Maleate Tablets; Drug: Capecitabine Tablets
- Arm G:JS105+Toripalimab Injection+Paclitaxel for Injection (Albumin Bound) (Experimental): JS105 administered orally, Toripalimab intravenous infusion, Paclitaxel (Albumin Bound) intravenous infusion
  Interventions: Drug: JS105; Drug: Toripalimab Injection; Drug: Paclitaxel for Injection (Albumin Bound)

INTERVENTIONS:
Drug: JS105 — JS105 is administered once daily, orally
Drug: Fulvestrant injection — Fulvestrant intramuscularly,The first cycle was injected once in D1 and D15, and then once in each cycle D1, and 28 days was 1 cycle
  Arms: Arm A:JS105+Fulvestrant Injection; Arm B:JS105+Fulvestrant Injection+Dalpiciclib Isetionate Tablets
Drug: Dalpiciclib Isetionate Tablets — Dalpiciclib Isetionate Tablets, QD, oral, taken continuously for 21 days, then stopped for 7 days, 28 days for a cycle
  Arms: Arm B:JS105+Fulvestrant Injection+Dalpiciclib Isetionate Tablets
Drug: Toripalimab Injection — Toripalimab Injection,Intravenous infusion, once every 3 weeks, 21 days for 1 cycle
  Arms: Arm C:JS105+Toripalimab Injection; Arm G:JS105+Toripalimab Injection+Paclitaxel for Injection (Albumin Bound)
Drug: Paclitaxel for Injection (Albumin Bound) — Paclitaxel for Injection (Albumin Bound),Intravenous infusion, D1, 8, 15 infusion, every 28 days for a cycle
  Arms: Arm D:JS105+Paclitaxel for Injection (Albumin Bound); Arm G:JS105+Toripalimab Injection+Paclitaxel for Injection (Albumin Bound)
Drug: Fluzoparib Capsules — Fluzoparib Capsules is administered once daily, orally
  Arms: Arm E:JS105+Fluzoparib Capsules
Drug: Pyrotinib Maleate Tablets — Pyrotinib Maleate Tablets is administered once daily, orally
  Arms: Arm F:JS105+Pyrotinib Maleate Tablets+Capecitabine Tablets
Drug: Capecitabine Tablets — Capecitabine Tablets is administered once daily, orally
  Arms: Arm F:JS105+Pyrotinib Maleate Tablets+Capecitabine Tablets

SUMMARY:
This study is an open-label, multicenter, Phase Ib/II clinical study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of JS105 in combination with other anti-tumor therapies in patients with advanced solid tumors. Patients will be enrolled in two stages: a dose-escalation stage and a dose-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form;
2. 18≤ age ≤ 75 years old, male or female;
3. Arms A and B, including the Dose Escalation Phase (Phase Ib) and Cohort Expansion Phase (Phase II):

   * Patients with histologically or cytologically confirmed recurrent/metastatic HR-positive and HER2-negative breast cancer;
   * HER2 negative must meet one of the following: IHC 0, IHC 1+; IHC2+ should be further confirmed by in situ hybridization (ISH) to determine HER2 negative, and different tissue blocks can also be selected for re-testing;
   * ER-positive and/or PR-positive: ER-positive requires >10% of tumor cell nuclei in the whole section to express ER;
   * For females, either postmenopausal or premenopausal/perimenopausal can be enrolled: postmenopausal, defined as meeting at least one of the following criteria: 1) age ≥ 60 years, 2) age < 60 years, and amenorrhea ≥ 12 months, and follicle-stimulating hormone and estradiol levels in the postmenopausal range in the absence of chemotherapy, endocrine therapy, or ovarian function suppression therapy, 3) prior bilateral oophorectomy. Premenopausal or perimenopausal (i.e., does not meet postmenopausal criteria) and meets the following criteria: Started at least 2 weeks before the first dose of study drug and continuously treated with luteinizing hormone-releasing hormone (LHRH) agonists (e.g., goserelin or leuprolide) for the duration of study treatment
   * For stage Ib, the patient has disease progression during or after prior endocrine therapy or other systemic therapy, with no limit on the number of prior lines of therapy;
   * For Group A Phase II, patients meet the following criteria: disease progression or recurrence during or after prior treatment with AI with or without CDK4/6 inhibitors, ≤2 lines of systemic therapy in advanced breast cancer, ≤1 line of chemotherapy (neoadjuvant/adjuvant chemotherapy is not counted as a line of chemotherapy), and > after completion of (neo)adjuvant endocrine therapy patients with recurrence at 12 months must receive 1 to 2 lines of systemic therapy for advanced disease to be enrolled;
   * For Group B stage II, patients who meet: recurrence during or ≤ 12 months after completion of (neo)adjuvant endocrine therapy or disease progression after receiving 1st line of endocrine therapy in the advanced stage, ≤ 1st line chemotherapy in the advanced breast cancer stage are allowed;
4. Arm C, including the Dose Escalation Phase (Phase Ib) and Cohort Expansion Phase (Phase II):

   * Patients with histologically or cytologically confirmed recurrent/metastatic endometrial and cervical cancer;
   * Disease progression or intolerance to standard therapy after receiving ≥1 line of systemic therapy;
5. Group D, including the Dose Escalation Phase (Phase Ib) and Cohort Expansion Phase (Phase II):

   ■ Patients with histologically or cytologically confirmed recurrent/metastatic triple-negative breast cancer or patients with advanced gynecologic tumors (including patients with epithelial ovarian, fallopian tube or primary peritoneal cancer, endometrial cancer, and cervical cancer);
   * Disease progression or intolerance to standard therapy after receiving ≥1 line of systemic therapy;
   * For stage II, in the case of ovarian cancer, must be a platinum-resistant/platinum-refractory patient (defined as disease progression during or within 6 months of completion of platinum-containing chemotherapy) For groups A, B, and D, stage Ib can be enrolled regardless of whether PIK3CA is mutated or not, and stage II should have PIK3CA activating mutations, which are determined by the central laboratory to be PIK3CA activating mutations by the sponsor. The test results of the preferred tissue sample are used as the basis for enrollment, and for patients who are truly unable to provide a tissue sample that meets the requirements, a positive PIK3CA mutation of the ctDNA test is allowed as the basis for enrollment.
6. Arm E, including the Dose Escalation Phase (Phase Ib) and Cohort Expansion Phase (Phase II):

   * Patients with histologically or cytologically confirmed recurrent/metastatic triple-negative breast cancer or epithelial ovarian, fallopian tube, or primary peritoneal cancer
   * Disease progression or intolerance to standard therapy after receiving ≥1 line of systemic therapy
   * For stage II, in the case of ovarian cancer, must be a platinum-resistant/platinum-refractory patient (defined as disease progression during or within 6 months of completion of platinum-containing chemotherapy)
7. Arm F, including the Dose Escalation Phase (Phase Ib) and Cohort Expansion Phase (Phase II):

   ■ Patients with histologically or cytologically confirmed recurrent/metastatic HER2-positive breast cancer;

   ■ Disease progression or intolerance to standard therapy after receiving ≥1 line of anti-HER2 therapy;
8. Group G: including Dose Escalation Phase (Phase Ib) and Cohort Expansion Phase (Phase II):

   * Patients with histologically or cytologically confirmed triple-negative breast cancer, i.e., HER2, ER, PR are all negative;
   * Patients with first-diagnosed stage IV (AJCC 8th edition) or recurrent/metastatic triple-negative breast cancer who are not candidates for surgical treatment, and have not received prior systemic therapy for advanced disease;
9. Agree to provide tumor tissue and blood samples for PIK3CA mutation testing required for enrollment:

   ■Tumor tissue specimens: fresh or archival unstained sections, preferably from tumor samples collected after the most recent disease progression or recurrence. Formalin-fixed, paraffin-embedded (FFPE) unstained sections (at least 5 surgical samples and 10 needle biopsy samples are recommended) are required. For patients who are unable to provide tissue samples or the number of sections is insufficient, it is necessary to communicate with the sponsor whether they can be enrolled;

   ■Freshly collected pre-treatment blood sample of at least 10ml
10. All acute toxicities due to prior antineoplastic therapy, surgery, or radiotherapy, etc., resolved to Grade 0-1 (according to NCI CTCAE version 5.0) or the level specified by the enrollment/exclusion criteria. Except for alopecia, pigmentation, or other toxicities that, in the opinion of the investigator, do not pose a safety risk to the patient and do not affect treatment compliance;
11. At least one measurable lesion (only for Phase II cohort expansion phase) or non-measurable osteolytic or mixed bone lesion (for breast cancer patients only) that meets the requirements of RECIST v1.1;
12. Eastern Cooperative Oncology (ECOG) performance status score: 0 or 1;
13. Expected survival ≥ 12 weeks;
14. Ability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening, or otherwise altering the dosage form of the product;
15. Functions of vital organs, in line with the requirements:

    a. No blood transfusion blood products or hematopoietic growth factors to correct the blood cell count within 14 days before the examination creatinine clearance was calculated using the Cockcroft/Gault formula: Creatinine clearance (mL/min) = (140-age)× Body weight (kg) ×(0.85 [females only]) 72 × serum creatinine (mg/dl) c. For patients with FPG ≥ 100 mg/dL and/or HbA1c ≥ 5.7% (eg, prediabetes threshold) during the screening period, lifestyle changes such as dietary prescription (eg, small and frequent meals, low-carb diet, high-fiber diet, etc.) and exercise are recommended according to ADA guidelines, and endocrinologist consultation is recommended.

    d. Patients receiving anticoagulant therapy (such as low molecular weight heparin or warfarin) should be stable at the dose of anticoagulant drugs for at least 4 weeks without dose adjustment; e. Only urine routine showed urine protein ≥2+, and additional 24-hour urine protein quantification was required
16. Within 7 days before the first dose of study drug, females of childbearing potential must confirm that the serum HCG test is negative and non-lactating, and female patients, as well as male patients whose partner is a female of childbearing age, need to use highly effective contraception during study treatment and within 30 days after the last dose of JS105 or during the contraceptive period specified in the label of other antineoplastic drugs, whichever occurs later, (see section 10.3 for the definition of WOCBP);

Exclusion Criteria:

1. Prior treatment with PI3K/AKT/mTOR inhibitors, prior treatment with fulvestrant and other SERDs (applicable to phase II of group A and phase II of group B);
2. Patients with known hypersensitivity to JS105 and/or the corresponding group of combination drug components;
3. Received the following treatments before the first dose of the study drug:

1) Major surgery or radiotherapy within 4 weeks, or anticipated major surgery (except tumor biopsy) or radiotherapy during the study; 2) Systemic chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin; oral fluorouracil can be shortened to 2 weeks or 5 half-lives of the drug, whichever is longer), targeted therapy (small molecule targeted drugs can be shortened to 2 weeks or 5 half-lives of the drug, whichever is longer), immunotherapy or biological therapy; 3) Receiving endocrine therapy or proprietary Chinese medicine preparations with anti-tumor indications within 2 weeks.

4) Other clinical investigational drugs (without placebo) within 4 weeks; 5) Vaccination with live attenuated vaccine within 4 weeks; 6) Received drug treatment with a known strong inhibitor or inducer of the isoenzyme CYP3A4 within 7 days (see Appendix 4 for a strong inhibitor or inducer of the isoenzyme CYP3A4); 7) Need for long-term use or use of ≥10mg/day prednisone and equivalent doses of systemic corticosteroids or immunosuppressive drugs within 2 weeks before the first dose; 4. Previous allogeneic bone marrow transplantation or solid organ transplantation; 5. Other malignancies other than study disease within 5 years before the first dose, except for malignancies that can be expected to heal after treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with radical surgery); 6. Patients with symptomatic, untreated, or ongoing central nervous system metastases requiring ongoing treatment (previously treated patients who have been stable for at least 3 months, have no disease progression as determined by imaging within 4 weeks before the first dose of the study, and all neurological symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and have stopped using radiation, surgery, or steroids at least 4 weeks before the first dose of study treatment, may be enrolled); 7. Pleural effusion, pericardial effusion, or ascites effusion (once a month or more frequent) that is uncontrolled or requires repeated drainage. Patients who need to be stable for at least 1 week before enrollment after drainage can be enrolled (stable is defined as no clear increase in pleural effusion without any intervention); 8. Concomitant and uncontrollable concomitant diseases, including but not limited to:

1. History of acute pancreatitis, history of chronic pancreatitis, or presence of pancreatic metastases within one year before screening;
2. Presence of type I diabetes mellitus or history of uncontrolled type II diabetes;
3. Ongoing active infection, unexplained fever > 38.5°C
4. Severe cardiovascular disease, including but not limited to a history of stroke or transient ischemic attack, angina pectoris, or myocardial infarction within 6 months before the first dose of study treatment, documented history of congestive heart failure (New York Heart Association Class II-IV) or cardiomyopathy, uncontrolled cardiac arrhythmia, active ventricular arrhythmia requiring medication or related history, symptomatic coronary heart disease or unstable angina;
5. History of interstitial pneumonia, drug-induced pneumonia, radiation pneumonitis requiring steroid treatment, or active pneumonitis with clinical symptoms, or other moderate to severe lung diseases that seriously affect lung function;
6. Presence of gastrointestinal insufficiency or gastrointestinal disease that may affect the swallowing (taking) or absorption of the study drug (e.g., ulcerative disease, uncontrolled vomiting, diarrhea, malabsorption syndrome, small bowel resection, history of active inflammatory bowel disease (such as Crohn's disease or ulcerative colitis), etc.); 9. Known human immunodeficiency virus (HIV) positive patient or active hepatitis B or C, except for the following:

1) Hepatitis B core antibody (HBcAb) positive and hepatitis B surface antigen (HBsAg) negative during the screening period can participate in this study; 2) Patients who are HBsAg positive and whose HBV DNA is less than the lower limit of detection can be enrolled, and the risk will be assessed by the investigator, if necessary, anti-HBV therapy should be received throughout the study treatment period to avoid viral activation; 3) Patients with positive HCV antibody can only be enrolled if the HCV RNA PCR test result is negative; 10. Female patients who are pregnant, lactating, or intend to become pregnant during the study; 11. Any other clinically significant disease or condition that, in the opinion of the investigator, could affect protocol compliance (such as a history of psychiatric illness or substance abuse), or affect the patient's signing of informed consent (such as drug use and substance abuse), or would be inappropriate to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | At the end of Cycle 1 (each cycle is 28 days)
  Incidence and severity of DLT events.
MTD | At the end of Cycle 1 (each cycle is 28 days)
  Maximum tolerated dose
RP2D | At the end of Cycle 1 (each cycle is 28 days)
  Recommended phase II dose
Incidence and severity of adverse events including serious adverse events | Up to 2 years
  Abnormal changes in clinical symptoms, vital signs, physical examination, laboratory tests, electrocardiograph and other examinations.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  Objective Response Rate (ORR) as Assessed by Investigator according to RECIST v1.1
Duration of Objective Response (DOR) | Up to 2 years
  Duration of Objective Response (DOR) as Assessed by Investigator according to RECIST v1.1
Disease Control Rate(DCR) | Up to 2 years
  Disease Control Rate(DCR)
Progression-Free Survival (PFS) | Up to 2 years
  Progression-Free Survival (PFS) as Determined by Investigator according to RECIST v1.1
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS)
AUC of JS105,dalpiciclib and fluzoparib | At pre-defined intervals up to 2 years
  Area under the curve of JS105,dalpiciclib and fluzoparib
Tmax of JS105, dalpiciclib and fluzoparib | At pre-defined intervals up to 2 years
  Time to reach maximum concentration of JS105,dalpiciclib and fluzoparib
Cmax of JS105,dalpiciclib and fluzoparib | At pre-defined intervals up to 2 years
  Maximum Plasma Concentration (Cmax) of JS105, dalpiciclib and fluzoparib
Vz/F of JS105, dalpiciclib and fluzoparib | At pre-defined intervals up to 2 years
  Apparent volume of distribution of JS105, dalpiciclib and fluzoparib
Clearance(CL) of JS105, dalpiciclib and fluzoparib | At pre-defined intervals up to 2 years
  Clearance(CL) of JS105, dalpiciclib and fluzoparib
Half-life(T1/2) of JS105, dalpiciclib and fluzoparib | At pre-defined intervals up to 2 years
  Half-life(T1/2) of JS105, dalpiciclib and fluzoparib

OTHER OUTCOMES:
The proportion of patients with PIK3CA mutations in tumor remission | Up to 2 years
  The proportion of patients with PIK3CA mutations in tumor remission

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No